CLINICAL TRIAL: NCT03640676
Title: Intermittent Negative Pressure to Improve Blood Flow in Patients With Peripheral Artery Disease: Effects After Long-term Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Otivio AS (Industry)
Responsible Party: Principal Investigator, Jonny Hisdal, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018/748
Record Dates: First submitted 2018-08-14; First posted 2018-08-21 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized sham-controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INP -10mmHg (Sham Comparator): In addition to standard medical treatment, patients will receive treatment with FlowOx, applying intermittent negative pressure of -10mmHg one hour in the morning and one hour in the evening at home for 12 weeks.
  Interventions: Device: FlowOx
- INP -40mmHg (Active Comparator): In addition to standard medical treatment, patient swill receive treatment with FlowOx, applying intermittent negative pressure of -40mmHg one hour in the morning and one hour in the evening at home for 12 weeks.
  Interventions: Device: FlowOx

INTERVENTIONS:
Device: FlowOx — FlowOx is a CE marked device developed to increase blood flow to the lower extremities. A pressure chamber is sealed around the leg below the knee and is connected to a control unit which induces pulses of 10 sec negative pressure, and 7 sec of atmospheric pressure.

SUMMARY:
Studies have shown that intermittent negative pressure (INP) can induce short-term increase in blood flow in the extremity in patients with peripheral artery disease (PAD). Case reports also have indicated that INP treatment has beneficial hemodynamic and clinical effects in patients with lower limb ischemia and hard to heal leg ulcers. However, the clinical and physiological effects of long-term INP treatment are not well documented and needs further investigation.

DETAILED DESCRIPTION:
A double-blinded randomized sham-controlled trial.

Otivio AS is the developer of FlowOx, a noninvasive CE marked device to increase blood flow to the lower extremity. The device acts as a pressure chamber sealed around the patient's lower leg, applying pulses of intermittent negative pressure and atmospheric pressure. The pressure pulses are generated by a control unit, alternating between removing air from- and venting the pressure chamber.

Preliminary tests indicate a significant increase in blood flow to the extremity during INP treatment at -40 mmHg, but a similar increase in blood flow was not detected during treatment INP treatment at -10 mmHg. Hence, treatment with -10 mmHg, may serve as a sham intervention, when evaluating the clinical and physiological effects of long-term INP treatment.

All patients will receive best medical treatment including advice for smoking cessation, dietary advice, and advice for physical exercise, and pharmacological treatment with statins and platelet inhibitors. Patients will be randomized into two groups, one group receiving INP treatment with a pressure of -10 mmHg, the other group receiving INP treatment with a pressure of -40 mmHg. Treatment will be conducted by the patient him/herself at home, one hour in the morning and one hour in the evening for 12 weeks.

Pain-free- and maximal walking distance, ankle-brachial index, arterial blood flow during application of INP, maximal blood flow, and biomarkers of inflammation and endothelial dysfunction will be registered at baseline and after 12 weeks to evaluate the effects of long-term INP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ankle-Brachial Index < 0,9, and intermittent claudication

Exclusion Criteria:

* Incapable to make an informed consent
* Inability to perform a treadmill test
* Inability to independently operate FlowOx
* Severe heart disease such as unstable angina pectoris, severe heart failure (NYHA IV), severe valve failure
* Severe COPD

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in maximal walking distance | At baseline and after 12 weeks of treatment
  Treadmill test
Change in pain-free walking distance | At baseline and after 12 weeks of treatment
  Treadmill test

SECONDARY OUTCOMES:
Change in serum levels of markers of inflammation and endothelial dysfunction | At baseline and after 12 weeks
  E-selectin, ICAM-I, IL1, IL-6, IL-8, TNF-alfa, TGF-beta, IL-10
Changes in resting and maximal blood flow | At baseline and after 12 weeks
  Strain-gauge plethysmography
Changes in Ankle-Brachial Index | At baseline and after 12 weeks
Changes in arterial blood flow during application of INP | At baseline and after 12 weeks
  Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Jonny Hisdal, PhD, Principal Investigator — Deprtment of Vascular Diseases, Oslo University Hospital
Locations (3):
- Norway (3):
  - Department of Surgery, Section of Vascular and Thoracic surgery, Sykehuset Sørlandet, Kristiansand
  - Department of Vascular Surgery, Oslo University Hospital, Aker, Oslo
  - Department of Vascular Surgery, St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoel H, Pettersen EM, Hoiseth LO, Mathiesen I, Seternes A, Seljeflot I, Hisdal J. Effects of intermittent negative pressure treatment on circulating vascular biomarkers in patients with intermittent claudication. Vasc Med. 2021 Oct;26(5):489-496. doi: 10.1177/1358863X211007933. Epub 2021 May 13. PMID 33985385